CLINICAL TRIAL: NCT05427825
Title: Anesthetic Protocols for Enhance Recovery After Metastatic Spine Tumor Resection Surgery: a Randomized Controlled Trial
Brief Title: ERAS Anesthetic Care for Metastatic Spine Cancer Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 202203092MINA
Record Dates: First submitted 2022-06-16; First posted 2022-06-22 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Metastatic Bone Tumor
MeSH Terms: conditions — Bone Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients in the treatment group received the study protocolized care bundle including multimodal anesthesia and HPI-assisted hemodynamic therapy.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS group (Experimental): Patients in the experimental group receive the protocolized anesthetic care bundle including EEG spectrum-guided multimodal anesthesia and HPI-guided hemodynamic therapy.
  Interventions: Other: ERAS anesthetic care
- Control (Active Comparator): Patients in the control group receive standard anesthetic care including bispetral index-guided balanced anesthesia and regular hemodynamic care protocols.
  Interventions: Other: Standard anesthetic care

INTERVENTIONS:
Other: ERAS anesthetic care — The ERAS anesthetic care includes EEG spectrum-guided multimodal anesthesia and HPI-guided hemodynamic therapy.
  Arms: ERAS group
Other: Standard anesthetic care — The standard anesthetic care includes bispectral index guided general anesthesia and arterial line monitored hemodynamic care.
  Arms: Control

SUMMARY:
Spinal metastases account for 60% of all malignant bone metastases and represent a medically important treatment goal. For patients with malignant tumors diagnosed at this stage, performing En bloc spondylectomy with wide margin of resection facilitate the improvement in quality of life including ambulatory ability, daily activities independence and attenuation of bone pain. However, En bloc spondylectomy is a major operation with long operation time and frequent hemodynamic instability during the operation. Therefore, the anesthetic care plays an important role and an enhanced recovery after surgery (ERAS) is the goal.

For the ERAS anesthesia protocol for En bloc spondylectomy, we propose two major components to achieve this goal: (1) an encephalographic spectrum guided multimodal anesthesia combined with ultrasound-guided nerve block and (2) the advanced machine-learning algorithm index, namely the hypotension predictive index (HPI) guided hemodynamic protocol.

DETAILED DESCRIPTION:
The anesthetic protocol comprises of two major proposed components to enhanced recovery after spine cancer total en bloc resection. First, a multimodal general anesthesia consisting of GABAnergic hypnotic agent (propofol or sevoflurane), ketamine and dexmedetomidine was conducted by using the encephalographic density spectrum array. In addition, ultrasound-guided erector spinae plane block is applied. These techniques potentially prevent anesthesia induced delirium and may profoundly improve postoperative analgesic quality. Second, advanced hemodynamic monitoring device, namely the hypotensio predictive index, will be used for prevention of intraoperative hypotension and facilitate precise transfusion protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing metastatic spine cancer resection surgery

Exclusion Criteria:

* Expected survival less than 6 months
* Previous surgery or radiotherapy for the spine metastasis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative quality of recovery-15 score (QoR-15) | 3 days
  Comparing the quality of recovery-15 score (0-150) at the first and third postoperative days

SECONDARY OUTCOMES:
Delirium incidence | 3 days
  Delirium diagnosed based on the Confusion Assessment Method (CAM) criteria during three days after surgery
Pain intensity | 3 days
  Postoperative pain intensity measure by using the visual analogue scale (0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Yu Wu, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan